CLINICAL TRIAL: NCT04226027
Title: Dynamically Tailoring Interventions for Problem-Solving in Diabetes Self-Management Using Self-Monitoring Data - a Randomized Controlled Trial (RCT)
Brief Title: Dynamically Tailored Behavioral Interventions in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Clinical Directors Network (Network); University of Colorado, Denver (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Olena Mamykina, PhD, Associate Professor of Biomedical Informatics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAS5528; R01DK113189 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Mobile health; Mhealth; T2.coach; Smartphone app
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm RCT with 1:1 randomization at participant level, with stratified randomization to balance by clinical site, sex, and language, evaluate the efficacy of the T2.coach intervention
Masking Description: Because of the nature of the intervention (smartphone app), masking is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2.coach (Experimental): Participants receive standard care (diabetes self-management education provided by their Federally Qualified Community Health Center) and are asked to use T2.coach for 6 months.
  Interventions: Behavioral: T2.coach
- Control (No Intervention): Participants receive standard care (diabetes self-management education provided by their Federally Qualified Community Health Center).

INTERVENTIONS:
Behavioral: T2.coach — T2.coach is a smartphone app for low-burden capture of diet and blood glucose (BG) levels and for reviewing past records, integrated with FitBit for captured of physical activity and sleep. All captured data are sent to the computational inference engine that uses machine learning methods and expert system to formulate personalized behavioral goals. Examples of behavioral goals include the following: "For high carbohydrate breakfasts, reduce your carbs to be about 1 carb choice. Examples of 1 carb choice are 1 slice of whole wheat toast, 1 cup of oatmeal, or 1 apple." The T2.coach chatbot companion uses text messages to help individuals set goals that are consistent with evidence based guidelines for diabetes self-management, inferences on data captured with T2.coach, and their own preferences, as well as send individuals goal reminders and prompts for reflection on goal achievement.
  Arms: T2.coach

SUMMARY:
In this project, the investigators will evaluate the efficacy of a novel approach to personalizing behavioral interventions for self-management of type 2 diabetes (T2DM) to individuals' behavioral and glycemic profiles discovered using computational learning and self-monitoring data. This study is a two-arm randomized controlled trial with n=280 participants recruited from the participating Federally Qualified Health Centers (FQHCs). The participants will be randomly assigned to the intervention group and the usual care (control) group with 1-1 allocation ratio. Half of the participants (n=140) will be randomly assigned to a usual care (control) group. Both groups will receive standard diabetes education at their respective FQHC site. In addition, the experimental group will receive instructions to use T2.coach for a minimum of 6 months.

DETAILED DESCRIPTION:
One of the main difficulties in managing diabetes is that each affected individual requires personally tailored combination of diet, exercise, and medication to effectively control their blood sugar. Rather than strictly following a doctor's prescription, individuals need to carefully examine their lifestyle choices and their impact on their health. Independent learning, experimentation and problem solving become of great importance. However, they can be challenging for individuals with diabetes. In this project, the investigators will refine and evaluate a novel intervention for diabetes self-management that uses computational analysis of self-monitoring data to help individuals with type 2 diabetes identify what daily activities, including consumption of meals, physical activity, and sleep, have impact on blood glucose levels, and suggest modifications to these daily activities to improve blood glucose levels.

Growing evidence highlights significant differences in glycemic function and cultural, social, and economical circumstances of individuals with type 2 diabetes (T2DM) that impact their self-management. Precision medicine strives to personalize medical treatment to an individual's genetic makeup, computationally discovered clinical phenotypes and lifestyle. Studies showed the benefits of tailoring not only medical treatment, but also behavioral interventions. Yet, currently, personalization of self-management in T2DM requires each individual to engage in discovery, reflection, and problem-solving-critical but cognitively demanding activities-or to rely on their healthcare providers. Both of these may present considerable barriers to individuals from medically under-served low income communities. Mobile health (mHealth) solutions in T2DM bring promise of reaching wider populations in need of self-management; however, few such solutions provide assistance with personalizing self-management behaviors. Ongoing efforts on personalizing behavioral interventions outside of T2DM focus on tailoring behavior modification techniques to individuals' psycho-social characteristics, such as self-efficacy ), and tailoring delivery of intervention to individuals' context rather than on personalizing self-management strategies.

The ongoing focus of this research is on developing informatics interventions for diabetes self-management, with a specific focus on discovery with self-monitoring data and on problem-solving for improving glycemic control. In the proposed research the investigators introduce T2.coach, an mHealth intervention that uses computational analysis of self-monitoring data to identify behavioral patterns associated with poor glycemic control and formulate personalized behavioral goals for changing problematic behaviors. This study will evaluate T2.coach's efficacy in a two-arm RCT with stratified randomization conducted with Clinical Directors Network (CDN), a well-recognized primary care practice-based research network (PBRN) of Federally Qualified Health Centers (FQHCs), and Agency for Healthcare Research and Quality (AHRQ)-designated Center of Excellence (P30) for Practice-based Research and Learning.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the health center for ≥ 6 months and a diagnosis of T2DM
* HbA1c ≥ 8.0,
* Aged 18 to 65 years
* Attends diabetes education program at the health center
* Owns a basic mobile phone
* Proficient in either English or Spanish

Exclusion Criteria:

* Pregnant
* Presence of severe cognitive impairment (recorded in patient chart),
* Existence of other serious illnesses (e.g. cancer diagnosis with active treatment, advanced stage heart failure, dialysis, multiple sclerosis, advanced retinopathy, recorded in patient chart),
* Plans for leaving the FQHC in the next 12 months,
* Participation in the previous trial of diabetes self-management technologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c value | Baseline, 6 months, 12 months
  Hemoglobin A1c

SECONDARY OUTCOMES:
DPSI Score | Baseline, 6 months, 12 months
  Diabetes Problem-Solving Inventory (DPSI) is a 9-item, open-ended questionnaire. Answers are coded on a Likert 5-point scale (1-very poor strategy; 5-excellent strategy). The final score ranges from 1 (lowest) to 5 (highest) and an overall score ≤3 indicates poor diabetes problem solving, so a higher score indicates a better outcome.
SCA-I Score | Baseline, 6 months, 12 months
  Diabetes Self-Care Inventory (SCA-I) is a 15-item 5-point Likert scale (1-never engage; 5-always engage) for measuring different aspects of diabetes self-care. The final score ranges from 1 (lowest) to 5 (highest) with a higher score indicating better self-care (better outcome).
DSES Score | Baseline, 6 months, 12 months
  Diabetes Self-Efficacy Scale (DSES) is a 15-item 10-point Likert scale (1-not at all confident; 4-totally confident) that measures the belief that one can self-manage one's own health, adapted to diabetes. The final score ranges from 1 (lowest) to 4 (highest) with a lower score indicating poor self-efficacy (worse outcome).
PAID Score | Baseline, 6 months, 12 months
  Problem Areas in Diabetes (PAID) is a 20-item 5-point Likert scale (0-not a problem; 4-very serious problem) that measures the emotional aspect of living with diabetes. The final score ranges from 0 (lowest) to 80 (highest), with a higher score indicating greater emotional discomfort (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Olena Mamykina, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Clinical Directors Network, New York, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of individual participant data (IPD) collected in this study, the dataset will only be made available for other potential users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.